CLINICAL TRIAL: NCT01706328
Title: A 12-Week Study to Evaluate the 24-Hour Pulmonary Function Profile of Fluticasone Furoate/Vilanterol (FF/VI) Inhalation Powder 100/25 mcg Once Daily Compared With Fluticasone Propionate/Salmeterol Inhalation Powder 250/50 mcg Twice Daily in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Study to Assess the Efficacy of Fluticasone Furoate/Vilanterol (FF/VI) Inhalation Powder 100/25 mcg Once Daily Compared With Fluticasone Propionate/Salmeterol Inhalation Powder 250/50 mcg Twice Daily in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116974
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Vilanterol (VI); Novel Dry Powder Inhaler (NDPI); FEV1; Fluticasone Furoate (FF); COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Albuterol; Health Services Needs and Demand

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FF/VI Inhalation Powder NDPI (Experimental): Subjects randomized to the FF/VI 100/25 arm will take an active inhalation of study medication during their morning dosing from their NDPI and will have an inhalation of dummy medication (placebo) as their morning ACCUHALER/DISKUS dose and as their evening dose.
  Interventions: Drug: FF/VI 100/25 Inhalation Powder NDPI; Drug: Placebo Inhalation Powder ACCUHALER/DISKUS; Drug: Salbutamol as needed
- Fluticasone Propionate/Salmeterol Inhalation Powder (Active Comparator): Subjects randomized to the Fluticasone Propionate/Salmeterol Inhalation Powder 250/50mcg arm will have an active dose of medication during both their morning and evening treatments from the ACCUHALER/DISKUS and a dummy placebo dose in the morning from their NDPI.
  Interventions: Drug: Fluticasone Propionate/Salmeterol 250/50 Inhalation Powder ACCUHALER/DISKUS; Drug: Placebo Inhalation Powder NDPI; Drug: Salbutamol as needed

INTERVENTIONS:
Drug: FF/VI 100/25 Inhalation Powder NDPI — Subjects randomized to the FF/VI Inhalation Powder Novel Dry Powder Inhaler (NDPI) arm will receive a single inhalation of 100 mcg FF and 25 mcg VI via NDPI every morning for 12 weeks.
  Arms: FF/VI Inhalation Powder NDPI
Drug: Fluticasone Propionate/Salmeterol 250/50 Inhalation Powder ACCUHALER/DISKUS — Subjects randomized to the Fluticasone Propionate/Salmeterol Inhalation Powder ACCUHALER/DISKUS arm will receive a single inhalation of 250 mcg Fluticasone Propionate and 50 mcg Salmeterol via ACCUHALER/DISKUS once in the morning and once in the evening for 12 weeks.
  Other Names: ACCUHALER and DISKUS are registered trade marks of the GlaxoSmithKline Group of companies
  Arms: Fluticasone Propionate/Salmeterol Inhalation Powder
Drug: Placebo Inhalation Powder NDPI — Subjects randomized to the Fluticasone Propionate/Salmeterol Inhalation Powder ACCUHALER/DISKUS arm will receive a single inhalation of placebo inhalation powder via NDPI every morning for 12 weeks.
  Other Names: ACCUHALER and DISKUS are registered trade marks of the GlaxoSmithKline Group of companies
  Arms: Fluticasone Propionate/Salmeterol Inhalation Powder
Drug: Placebo Inhalation Powder ACCUHALER/DISKUS — Subjects randomized to the FF/VI Inhalation Powder NDPI arm will receive a single inhalation of placebo inhalation powder via ACCUHALER/DISKUS once in the morning and once in the evening for 12 weeks.
  Arms: FF/VI Inhalation Powder NDPI
Drug: Salbutamol as needed — Salbutamol inhalation powder

SUMMARY:
This will be a Phase IIIb multicentre, randomized, double-blind, double-dummy, 12-week parallel group study evaluating the effects of once daily in the morning treatment of FF/VI Inhalation Powder versus Fluticasone Propionate/Salmeterol Inhalation Powder twice daily on lung function in COPD subjects.

Subjects will be screened and will enter a 2-week, single-blind (placebo), Run-In Period to evaluate the subject's adherence with study treatment, study procedures and assessment of disease stability.

At the end of the Run-In Period, subjects will return to the Clinic and who meet all of the Randomization Criteria will be randomized to double-blind study medication (12-week treatment period). Subjects will be randomized to receive either FF/VI 100/25 via NDPI or Fluticasone Propionate/Salmeterol 250/50mcg via ACCUHALER/DISKUS. Matching placebos will be available in NDPI and ACCUHALER/DISKUS. Each morning (approximately 6-10 AM) subjects will take 1 inhalation from the NDPI followed by 1 inhalation from the ACCUHALER/DISKUS. Each evening (approximately 6-10 PM), approximately 12 hours after the morning dose with blinded study medication, subjects will take 1 inhalation from the ACCUHALER/DISKUS. Subjects will return to the clinic at the end of the treatment period.

A follow-up phone contact will be performed approximately 7 days after the last clinic visit. The overall study duration (Screening to Follow-up) for each subject is approximately 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A male or female >=40 years of age at Screening (Visit 1).
* Capable of giving written informed consent.
* Female subjects must be post-menopausal or using a highly effective method for avoidance of pregnancy.
* Subjects with a clinical history of COPD in accordance with the following definition by the American Thoracic Society/European Respiratory Society.
* Subject with a measured post-albuterol (salbutamol) FEV1/forced vital capacity(FVC) ratio of <=0.70 at Screening.
* Subjects with a measured post-albuterol (salbutamol) FEV1 <=70% of predicted normal values.
* Subjects with a current or prior history of ≥10 pack-years of cigarette smoking at Screening.

Exclusion Criteria:

* Current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD).
* Other respiratory disorders (alpha1-antitrypsin deficiency as the underlying cause of COPD, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, pulmonary fibrosis, pulmonary hypertension, interstitial lung diseases, or other active pulmonary diseases).
* Lung volume reduction surgery within the 12 months prior to Screening.
* Hospitalized due to poorly controlled COPD within 12 weeks of Screening.
* Poorly controlled COPD (occurrence of the following in the 6 weeks prior to Screening -Acute worsening of COPD that is managed by the subject with corticosteroids or antibiotics or that requires treatment prescribed by a physician).
* Lower respiratory tract infection that required the use of antibiotics within 6 weeks prior to Screening.
* Moderate/severe COPD exacerbation/lower respiratory tract infection during Run-In Period.
* Abnormal and clinically significant 12-lead ECG at Screening
* Historical or current evidence of uncontrolled or clinically significant disease like cardiovascular, hypertension, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease), peptic ulcer disease, or haematological abnormalities. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* History of hypersensitivity to any of the study medications or components of the inhalation powder; or history of severe milk protein allergy.
* Known or suspected history of alcohol or drug abuse within the last 2 years.
* Subjects who are medically unable to withhold their albuterol (salbutamol) and/or their ipratropium for the 4-hour period required prior to spirometry testing at each study visit.
* The subject has taken any other investigational drug within 30 days or 5 half-lives of the investigational product (IP) prior to the first dosing day in the current study.
* Use of additional medications prior to Screening (list of medications and time intervals are different for different class of medications and are indicated in the protocol)
* Subjects receiving treatment with long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day. Oxygen prn use (i.e., <=12 hours per day) is not exclusionary.
* Subjects who have participated in the acute phase of a Pulmonary Rehabilitation Program within 4 weeks prior to Screening
* Subjects at risk of non-compliance, or unable to comply with study procedures.
* Study investigators, sub-investigators, study coordinators, employees of a participating investigator or immediate family members of the aforementioned are excluded from participating in this study.
* Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Previously randomized to either the HZC113109 or HZC112352 clinical studies.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 828 (Actual)
Dates: Start 2012-10-15 (Actual); Primary Completion 2013-06-17 (Actual); Study Completion 2013-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (49):
- United States (16):
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Woodbury, Minnesota
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Renton, Washington
- Germany (10):
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Romania (11):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Brăila
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Râmnicu Vâlcea
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Timișoara
- Russia (9):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Kursk
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Vladivostok
  - GSK Investigational Site, Yaroslavl
- Ukraine (3):
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Dransfield MT, Feldman G, Korenblat P, LaForce CF, Locantore N, Pistolesi M, Watkins ML, Crim C, Martinez FJ. Efficacy and safety of once-daily fluticasone furoate/vilanterol (100/25 mcg) versus twice-daily fluticasone propionate/salmeterol (250/50 mcg) in COPD patients. Respir Med. 2014 Aug;108(8):1171-9. doi: 10.1016/j.rmed.2014.05.008. Epub 2014 Jun 19. PMID 24998880
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 116974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116974 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only those participants that started the Double-blind Treatment Period were considered enrolled.
Pre-assignment Details: At Visit 1, participants entered a 2-week, single-blind (placebo) Run-in Period to obtain Baseline assessments of salbutamol use and to evaluate adherence with study treatment and procedures, diary card completion, and assessment of disease stability. At Visit 2, participants were randomized to a 12-week, double-blind Treatment Period.
Groups:
- Placebo + Salbutamol: Participants were instructed to take single-blind placebo twice a day (one inhalation from a multi-dose powder inhaler [MPI] and one inhalation from a dry powder inhaler [DPI] in the morning; one inhalation from an MPI in the evening). In addition, all participants received supplemental albuterol (salbutamol) (via a metered dose inhaler [MDI] and/or nebules) to be used on an as-needed basis. Ipratropium bromide alone was permitted, provided that the participant was on a stable dose from Visit 1 (Screening) and remained on the stable dose throughout the study; however, ipratropium must have been withheld for 4 hours prior to and during each clinic visit.
- FF/VI 100/25 µg QD: Participants received one inhalation of fluticasone furoate/vilanterol (FF/VI) 100/25 micrograms (µg) once daily (QD) in the morning from a DPI and placebo twice daily (BID) from a DPI (one inhalation in the morning and one inhalation in the evening) for 12 weeks. In addition, participants were provided supplemental albuterol (salbutamol) inhalation to be used as needed throughout the study.
- FP/Salmeterol 250/50 µg BID: Participants received fluticasone propionate (FP)/salmeterol 250/50 µg BID from a DPI (one inhalation in the morning and one inhalation in the evening) plus placebo QD in the morning from a DPI for 12 weeks. In addition, participants were provided supplemental albuterol (salbutamol) to be used as needed throughout the study.
Period: 2-week Run-in Period
Arm/Group | Placebo + Salbutamol | FF/VI 100/25 µg QD | FP/Salmeterol 250/50 µg BID
Started | 993 | 0 | 0
Completed | 828 | 0 | 0
Not Completed | 165 | 0 | 0
Not completed — Inclusion/Exclusion Criteria Not Met | 140 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Period: 12-week Double-blind Treatment Period
Arm/Group | Placebo + Salbutamol | FF/VI 100/25 µg QD | FP/Salmeterol 250/50 µg BID
Started | 0 | 412 | 416
Completed | 0 | 366 | 371
Not Completed | 0 | 46 | 45
Not completed — Adverse Event | 0 | 14 | 16
Not completed — Lack of Efficacy | 0 | 4 | 4
Not completed — Protocol Violation | 0 | 4 | 2
Not completed — Protocol-defined Stopping Criteria Met | 0 | 11 | 9
Not completed — Lost to Follow-up | 0 | 3 | 1
Not completed — Physician Decision | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FF/VI 100/25 µg QD | FP/Salmeterol 250/50 µg BID | Total
Number analyzed (Participants) | 412 | 416 | 828
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.0 (8.17) | 61.3 (8.37) | 61.1 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 122 | 233
  Male | 301 | 294 | 595
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 9 | 5 | 14
  American Indian or Alaska Native | 0 | 1 | 1
  White-White/Caucasian/European Heritage | 403 | 410 | 813

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Trough in Weighted-mean 24-hour Serial Forced Expiratory Volume in One Second (FEV1) on Treatment Day 84
Description: FEV1 is a measure of lung function and is defined as the volume of air that can be forcefully exhaled in one second. The weighted mean was calculated from the pre-dose FEV1 and the post-dose FEV1 measurements taken at 5, 15, 30, and 60 minutes and 2, 4, 6, 8, 12, 13, 14, 16, 20, and 24 hours on Treatment Day 84. Baseline trough FEV1 was calculated as the mean of the two assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1. The weighted mean was derived by calculating the area under curve, and then dividing by the relevant time interval. The weighted mean change from Baseline was calculated as the weighted mean of the 24-hour serial FEV1 measurements on Day 84 minus the Baseline trough FEV1 value. The analysis used an analysis of covariance (ANCOVA) model with covariates of Baseline FEV1, reversibility stratum, smoking status (at Screening), country, and treatment.
Time Frame: Baseline and Day 84
Population: Intent-to-Treat (ITT) Population: all participants who were randomized and received at least one dose of study drug. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF/VI 100/25 µg QD | FP/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 350 | 356
Liters | 0.168 (0.0121) | 0.142 (0.0120)
Statistical Analysis 1: Comparison: FF/VI 100/25 µg QD vs FP/Salmeterol 250/50 µg BID; Test type: Superiority or Other; p = 0.137, ANCOVA; Mean Difference (Net) = 0.025, 95% CI 2-sided [-0.008 to 0.059]

2. Secondary Outcome: Time to Onset on Treatment Day 1
Description: Time to onset on Treatment Day 1 is defined as the time to an increase of 100 milliliters (mL) from Baseline in FEV1 during the 0- to 4-hour serial measurements (5, 15, 30, 60, 120, and 240 minutes post-dose). Participants who never met or exceeded a 100 mL increase over the Baseline value during the 4-hour serial measurements were censored at the actual time of their last FEV1 measurement.
Time Frame: Baseline and Day 1
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Median (Full Range); unit: Minutes
Arm/Group | FF/VI 100/25 µg QD | FP/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 411 | 416
Minutes | 15 [5 to 240] | 15 [5 to 240]

3. Secondary Outcome: Change From Baseline in Trough FEV1 on Treatment Day 85
Description: FEV1 is a measure of lung function and is defined as the volume of air that can be forcefully exhaled in one second. Trough FEV1 is defined as the 24-hour FEV1 assessment, which was obtained on Day 85. Baseline trough was calculated as the mean of the two assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1. Change from Baseline was calculated as the average of the Day 85 values minus the Baseline value. The analysis used an analysis of covariance (ANCOVA) model with covariates of Baseline FEV1, reversibility stratum, smoking status (at Screening), country, and treatment.
Time Frame: Baseline and Day 85
Population: ITT Population. Only those participants available at the indicated time point were assessed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF/VI 100/25 µg QD | FP/Salmeterol 250/50 µg BID
Number analyzed (Participants) | 364 | 369
Liters | 0.151 (0.0126) | 0.121 (0.0125)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication until Follow-up (up to 12 weeks).
Description: SAEs and non-serious AEs were collected in members of the ITT Population, comprised of all participants who were randomized and received at least one dose of study drug.
Arm/Group | FF/VI 100/25 µg QD | FP/Salmeterol 250/50 µg BID
Serious Adverse Events (participants affected / at risk) | 13/412 | 20/416
Other Adverse Events (participants affected / at risk) | 46/412 | 52/416
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg QD (N=412) | FP/Salmeterol 250/50 µg BID (N=416)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 4
Infective exacerbation of chronic obstructive airways diseas (Infections and infestations) | 0 | 3
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg QD (N=412) | FP/Salmeterol 250/50 µg BID (N=416)
Nasopharyngitis (Infections and infestations) | 30 | 26
Headache (Nervous system disorders) | 18 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.